CLINICAL TRIAL: NCT07371039
Title: Effects of a Nurse-Led Sacral Pressure Intervention During Labor on Pain Perception and Maternal Satisfaction: A Randomized Controlled Trial
Brief Title: Sacral Pressure During Labor: Effects on Pain and Maternal Satisfaction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Kavram Vocational School (Other)
Responsible Party: Principal Investigator, Ayşegül Muslu, Lucturer (PhD), Izmir Kavram Vocational School
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: E1881
Record Dates: First submitted 2026-01-14; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Getting Pregnant; Labor Pain; Intrapartum Period; 37-42 Weeks of Gestation; Singleton Fetus; Aged 18 Years or Older
Keywords: pregnant; labor pain; intrapartum period; nursing practices; clinical intervention
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacral massage applied to the S4-S5 bones (Experimental): Pressure will be applied to minimize the mother's pain in order to facilitate contractions.
  Interventions: Other: manual pressure application
- routine clinical practice (No Intervention)

INTERVENTIONS:
Other: manual pressure application — Pressure application using the metacarpal bone of one hand on the S4-S5 bones was planned.
  Arms: Sacral massage applied to the S4-S5 bones

SUMMARY:
The study will be conducted with pregnant women in the active and transitional phases of labor. In the intervention group, sacral pressure will be applied during contractions, while the control group will receive routine clinical care. Perceived labor pain and maternal satisfaction will be assessed throughout the labor process

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Singleton pregnancy
* Cephalic (vertex) presentation
* Gestational age between 37 and 42 weeks

Exclusion Criteria

* Illiterate in Turkish
* Presence of chronic disease(s)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals who come to the delivery room to give birth will participate.
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
The VAS Pain Scale | Average: 1 year

SECONDARY OUTCOMES:
The Intrapartum Period Satisfaction Form | Average: 1 year

CONTACTS AND LOCATIONS:
Overall Officials: AYSEGÜL MUSLU, Principal Investigator — izmir kavram vocation

IPD SHARING:
Plan to Share IPD: No